CLINICAL TRIAL: NCT00449774
Title: An Open-label, Randomised, Single-dose, Parallel-group Study to Demonstrate Bioequivalence of Two Formulations and the Effect of Food and Water on One Formulation of Lamotrigine in Healthy Male and Female Volunteers
Brief Title: Bioequivalence And Effect Of Food And Water On Lamotrigine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBI108617
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Mental Disorders
Keywords: Food effect; Safety; Tolerability; Water effect; Bioequivalence
MeSH Terms: conditions — Mental Disorders | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects in Treatment regimen C (Experimental): Subjects in treatment regimen C will receive 200 milligram (mg) orally disintegrating tablets (ODT) of lamotrigine disintegrate in mouth without water in fasting condition.
  Interventions: Drug: Lamotrigine ODT tablets
- Subjects in Treatment regimen D (Experimental): Subjects in treatment regimen D will receive 200 mg Immediate Release (IR) tablets of lamotrigine with water in fasting condition.
  Interventions: Drug: Lamotrigine IR tablets
- Subjects in Treatment regimen E (Experimental): Subjects in treatment regimen E will receive 200 mg ODT disintegrate of lamotrigine in mouth without water in fed state.
  Interventions: Drug: Lamotrigine ODT tablets
- Subjects in Treatment regimen F (Experimental): Subjects in treatment regimen F will receive 200 mg ODT of lamotrigine, that subjects will swallow with water in fasting condition.
  Interventions: Drug: Lamotrigine ODT tablets

INTERVENTIONS:
Drug: Lamotrigine IR tablets — Lamotrigine IR tablets will be available in dose strength of 200 mg.
  Other Names: Lamotrigine
  Arms: Subjects in Treatment regimen D
Drug: Lamotrigine ODT tablets — Lamotrigine ODT tablets will be available in dose strength of 200 mg.
  Arms: Subjects in Treatment regimen C; Subjects in Treatment regimen E; Subjects in Treatment regimen F

SUMMARY:
This study intends to demonstrate bioequivalence of two formulations, the effect of food and water on one formulation and safety and tolerability of two formulations of lamotrigine in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 19 to 55 years inclusive
* BMI within the range 19 to 32 kg/m2 inclusive.

Exclusion Criteria:

* Female subjects of childbearing potential will not be eligible if they are unwilling or unable to use an appropriate method of contraception at least 30 days prior to the first study drug through 30 days.
* Female subject is pregnant or lactating.
* Female subjects using hormonal contraceptive precautions including progesterone-coated intra-uterine device (IUD).
* Female subjects using hormonal replacement therapy.
* History of regular alcohol consumption > 7 drinks week for women and 14 drinks week for men
* Current smokers of 10 or more cigarettes per day

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2007-05-07 (Actual); Primary Completion 2007-06-19 (Actual); Study Completion 2007-06-19 (Actual)

PRIMARY OUTCOMES:
Lamotrigine AUC(0-inf) and Cmax. Time points when measures are taken : 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours | Time points when measures are taken : 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours

SECONDARY OUTCOMES:
Serum lamotrigine AUC(0-t), tlag, tmax,lambdaZ and t1/2 at the times shown above. Adverse events, changes in biochemistry, haematology, urinalysis parameters, electrocardiogram parameters, blood pressure and heart rate at various times during the study. | Serum lamotrigine AUC(0-t), tlag, tmax,lambdaZ and t1/2 at the times shown above

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study LBI108617 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/LBI108617?search=study&search_terms=LBI108617#rs
- Available data/document: Individual Participant Data Set: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LBI108617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register